CLINICAL TRIAL: NCT06424470
Title: A Randomized, Double-blind, Placebo-controlled Phase III Clinical Study Evaluating the Efficacy and Safety of Stapokibart Injection in Subjects With Prurigo Nodularis
Brief Title: Study on the Treatment of Prurigo Nodularis With Stapokibart Injection
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM310-110201
Record Dates: First submitted 2024-05-16; First posted 2024-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Prurigo Nodularis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stapokibart (Experimental): Stapokibart Injection, subcutaneous injection (SC)
  Interventions: Biological: Stapokibart
- Placebo (Placebo Comparator): subcutaneous injection (SC)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Stapokibart — Stapokibart Injection
  Arms: Stapokibart
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is a multicenter, randomized, double-blind, placebo-controlled phase III clinical study to evaluate the efficacy and safety of Stapokibart Injection in the treatment of subjects with prurigo nodularis, and observe pharmacokinetic characteristics, pharmacological effects, and immunogenicity.

DETAILED DESCRIPTION:
Chronic prurigo (CPG) is an independent chronic inflammatory skin disease characterized by chronic itching and multiple local or systemic prurigo lesions. Prurigo nodularis (PN) is the main subtype of CPG.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and agree to comply with the experimental process of this study and voluntarily sign the informed consent form.
* 18 ≤ Age ≤ 75 years old.
* Received at least 2 weeks of moderate or more potent topical corticosteroid therapy with insufficient efficacy.

Exclusion Criteria:

* With drug-induced prurigo nodularis.
* With clinically significant diseases.
* With severe liver and kidney function damage at the screening.
* With malignant tumors within the first 5 years before the screening.
* Plan to undergo major surgical procedures during this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2024-06-25 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects improved by ≥ 4 points from baseline on the Worst Itch Numerical Rating Scale (WI-NRS) at week 24 of treatment. | Up to week 24
  The Worst Itch Numerical Rating Scale (WI-NR) is a patient-reported outcome (PRO) consisting of individual items with scores ranging from 0 ("no itching") to 10 ("the most severe itching imaginable"). Subjects are required to use this scale to rate the severity of their most severe itching in the past 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Xinghua Gao, Principal Investigator — First Hospital of China Medical University
Locations (1):
- The First Hospital of China Medical University, Shenyang, Liaoning, China